CLINICAL TRIAL: NCT06024395
Title: A Stepped-Care Approach to Treating Dental Fear: A Sequential, Multiple Assignment, Randomized Trial for Cognitive-Behavioral Treatment Via Mobile App and Evidence-Based Collaborative Care
Brief Title: A Stepped Care Approach to Treating Dental Fear
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: New York University (Other)
Collaborators: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Treatment
Other Study IDs: 23-042-E
Record Dates: First submitted 2023-08-21; First posted 2023-09-06 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-06

CONDITIONS: Dental Fear

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dental FearLess App (Experimental): Dental FearLess app is an e-health intervention that includes psychoeducation about anxiety; affective, cognitive, and behavioral strategies for coping at the dentist.
  Interventions: Behavioral: Dental FearLess
- Treatment as Usual (No Intervention)

INTERVENTIONS:
Behavioral: Dental FearLess — Dental FearLess is a self-administered CBT-based mobile app that takes approximately 1 hour to complete.
  Arms: Dental FearLess App

SUMMARY:
The purpose of this study is to compare an intervention for dental fear to the usual approach (i.e., whatever participants' dentist typically does to help participants manage their fear). The dental fear intervention has 2 separate steps. Step 1 (the less intensive or 'light touch' intervention step) involves using a mobile application (app). Step 2 consists of a one-hour telehealth session with a mental health provider tailored to individualized dental fear.

This is a randomized study. The time spent participating in the study will depend on which study condition(s) participants are randomly assigned to. Because this study compares the dental fear intervention to the standard approach, 25% of participants will not get the intervention during the study period. These participants (called controls) will be offered the opportunity to provide feedback about their experiences with dentists. Participants will be offered the intervention free of charge at the conclusion of the study.

For each step of the intervention (Dental FearLess app or one-on-one session) relative to treatment as usual, the investigators hypothesize that participants will show greater declines in self-reported dental fear and improved oral health-related quality of life at post-treatment and follow-up period. De-identified attendance records will be collected from dental practices.

ELIGIBILITY:
Inclusion Criteria:

* Provide signed and dated informed consent/ assent form
* Willing to comply with all study procedures and be available for the duration of the study
* Be least 13 years old.
* Score 4 or above on the Gatchel single-item dental fear rating scale
* Willingness to allow access to dental attendance records
* Access to a smartphone or tablet

Exclusion Criteria:

Given the scope and nature of the study, there is no exclusion criteria.

Ages: 13 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1250 (Estimated)
Dates: Start 2023-09-11 (Actual); Primary Completion 2028-04-30 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Reduction of moderate to severe dental fear. | baseline, upto 8 weeks, 5/6 month follow-up visit
  Assess the efficacy of a CBT-based stepped-care (i.e., progressive treatment dosing) approach in the reduction of moderate to severe dental fear (measured via subjective report on IDAF).

CONTACTS AND LOCATIONS:
Overall Officials: Richard Heyman, Ph.D, Principal Investigator — New York University; Mark Wolff, DDS, Principal Investigator — University of Pennsylvania
Locations (1):
- New York University, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No